CLINICAL TRIAL: NCT02571127
Title: Ph IV , Longitudinal, Prospective, Open Label, Non-comparative, to Evaluate the Efficacy, Safety and Tolerability of a Non-hormonal Intravaginal Gel in Postmenopausal Women With Symptoms of Vaginal Dryness.
Brief Title: Evaluate the Efficacy, Safety and Tolerability of a Non-hormonal Intravaginal Gel in Postmenopausal Women With Symptoms of Vaginal Dryness.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Farmoquimica S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hidra 1
Record Dates: First submitted 2015-09-01; First posted 2015-10-08 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-09

CONDITIONS: Vaginal Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Only treatment (Experimental): two weekly applications (monday and thursday or tuesday and friday) for 12 weeks
  Interventions: Drug: Hidra1

INTERVENTIONS:
Drug: Hidra1 — Parameters: Vaginal health index (VHI) : The parameter of efficiency : a vaginal moisture ; Will Measured through the VHI : 1 = none / inflamed area ; 2 = no / NOT inflamed surface ; 3 = minimal, 4 = moderate and 5 = normal.
  Will be described through the Media and Standard Deviation or median and interquartile rank , as Minimum and Maximum.
  Scala: pH tape: It will be measured by its own value. Questionnaire: Sexual Function Index female (FSFI): internationally validated questionnaire with single answers for patient.
  Other Names: Parameters: Vaginal health index (VHI); Scala: pH tape; Questionnaire: Sexual Function Index female (FSFI)

SUMMARY:
Primary: Evaluation of improved vaginal moisture in postmenopausal women.

Secondary: the improvement of symptoms resulting from the dryness Rating (VHI), evaluation of the decrease in vaginal pH, assessment of Sexual Function Index female (FSFI), evaluation of adherence to study treatment by patient diary, assessing the acceptability of the product and subjective assessment of the patient as the itching and stinging / burning, beyond the safety assessment.

DETAILED DESCRIPTION:
ENDPOINT:

* Primary: Evaluation of improved vaginal moisture in post menopausal women through vaginal health index (VHI);
* Secondaryevaluate the increase in fluid volume, vaginal elasticity and integrity of the epithelium by the VHI, evaluate the pH control, improvement of female sexual quality by applying the Sexual Function Index female (FSFI), evaluate through the patient's daily treatment adherence, evaluate the acceptability (welfare, run-off and satisfaction) of the product and the improvement of itching and stinging / burning through questionnaires and verify the tolerability and safety by identifying adverse events.

STUDY DESING: Phase IV study, longitudinal, prospective, open label, non-comparative

POPULATION: Forty-six (46) post menopausal women with vaginal dryness

DRUG: Polimers and Sodium Lactate

TREATMENT: Only treatment - two weekly applications (monday and thursday or tuesday and friday) for 12 weeks

EVALUATION: The evaluation of the effectiveness will be held on all visits by medical clinical evaluation, evaluation of symptoms resulting from the dryness (VHI), pH evaluation (pH tape) and evaluation of female sexual quality (FSFI) and subjective evaluation as well as the compliance through the patient diary. The evaluation of the acceptability of the product will be the last visit by a questionnaire. The safety assessment will be carried out on all visits by identifying adverse events

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 40 years.
* in healthy postmenopausal women (not menstruating for more than one year).
* Women with vaginal dryness (VHI score in item vaginal moisture between 1-3)
* women with active sex lives of at least one sexual intercourse in the month
* Women without a history of sensitivity to similar formulations.
* understanding and signing an informed consent agreement.

Exclusion Criteria:

* Women in using other intravaginal gel moisturizer.
* Women diagnosed with cancer.
* Women with disease or condition that, in the opinion of the gynecologist, could affect the test results.
* Women using hormone replacement therapy in the last 3 months.
* Absence of history or visible evidence of chronic skin disease or regional infections.
* Women with genital herpes, vaginal infections or urinary tract infection.
* Pregnant women and nursing mothers.
* Personal history of allergy and hypersensitivity to any product of feminine hygiene.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-02 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of improved vaginal moisture in post menopausal women by the Vaginal health index (VHI). | 4 months
  Vaginal health index (VHI) : The parameter of efficiency : a vaginal moisture ; Will Measured through the VHI : 1 = none / inflamed area ; 2 = no / NOT inflamed surface ; 3 = minimal, 4 = moderate and 5 = normal
Scala: pH tape: It will be measured by its own value. | 4 months
Questionnaire: Sexual Function Index female (FSFI): internationally validated questionnaire with single answers for patient. | 4 months

SECONDARY OUTCOMES:
Verify the tolerability and safety by identifying adverse events | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Thales Braga, Analist, Study Chair — Famorquimica SA